CLINICAL TRIAL: NCT01470573
Title: Regenerative Medicine in Ocular Surface: Application of Cell Therapy for Ocular Surface Repair Using Progenitor Autologous Cells of Sclerocorneal Limbus Amplified ex Vivo
Brief Title: Regenerative Medicine in Ocular Surface: Application of Cell Therapy for Ocular Surface Repair Using Progenitor Cells of Sclerocorneal Limbus Amplified ex Vivo
Acronym: MeRSO09
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Sara Varea, Clinical Research Manager, Fundacion Clinic per a la Recerca Biomédica
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MeRSO09
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Unilateral Limbic Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Progenitor Autologous Cells (Experimental): Progenitor Autologous Cells of Sclerocorneal Limbus Amplified ex Vivo
  Interventions: Procedure: biological replacement corneal surface

INTERVENTIONS:
Procedure: biological replacement corneal surface — the expanded tissue will be applied to patient to replace the damaged ocular surface

SUMMARY:
Progenitor limbo sclerocorneal cells have properties of proliferation and differentiation to corneal and conjunctival epithelium. This cells can be isolated and ex vivo expanded using cell culture technics that could permit the biological replacement of damaged ocular surface.

ELIGIBILITY:
principal Inclusion Criteria:

* Serious unilateral limbic insufficiency
* Normal ophthalmological clinical examination in the opposite eye (biopsied eye)

Exclusion Criteria:

* one-eyed
* serious disorders in palpebral dynamics
* bilateral limbic insufficiency, immunological, systemic or local illness like toxical epidermic necrosis or pemphigoid
* breastfeeding or pregnancy
* positive serology of HIV, VLTH, HVC, HVB, CMV, Trypanosoma Cruzi or Treponema Pallidum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 6 months
  visual acuity improvement

SECONDARY OUTCOMES:
Improvement in appearance of ocular surface | 6 months
  presence of corneal epithelium de novo
lack of scar tissue in ocular surface | 6 months
decrease of preexisting corneal vascularization | 6 months
Improvement of corneal transparency | 6 months
absence or decrease of corneal conjunctivalization | 6 months
  the amount of caliciform cells using impression cytology will be compare between screening and 6 months visit
adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo P Casaroli Marano, MD PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (3):
- Spain (3):
  - Instituto Universitario Barraquer, Barcelona, Barcelona
  - Instituto de Microcirugía Ocular, Barcelona, Barcelona
  - Hospital Clinic of Barcelona, Barcelona, Barcelona